CLINICAL TRIAL: NCT01390753
Title: Preventing Respiratory Disease Hospitalizations in Premature Infants Fed Donor Human Milk
Brief Title: Role of Human Milk Bank in the Protection of Severe Respiratory Disease in Very Low Birth Weight Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Infant (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INFANT-001; Donor milk study (Other Grant/Funding Number: Thrasher)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Preterm formula (No Intervention)
- Donor milk + preterm formula (Active Comparator): Human milk from a donor bank
  Interventions: Dietary Supplement: Human donor milk
- Breastfeeding + formula (No Intervention)
- Breasfeeding (No Intervention)

INTERVENTIONS:
Dietary Supplement: Human donor milk
  Arms: Donor milk + preterm formula

SUMMARY:
Acute respiratory infections are the leading cause of hospitalization in premature infants worldwide. Severity rates are particularly high in developing countries. Numerous viruses can cause severe disease, but the most frequent agent of hospitalization is respiratory syncytial virus (RSV). In a recent study in Argentina, 58% of RSV infected VLBW infants required hospitalization and 19% required mechanical ventilation. One every twenty infected infants died. Unlike industrialized nations, VLBW infants in developing countries often lack access to prophylaxis against RSV with a commercially available monoclonal antibody (palivizumab). No vaccine or preventive intervention is available against any respiratory virus for infants younger than 6 months of age in developing countries and the public sector of most middle-income countries.

The protective role of breastfeeding against respiratory infections in developing countries is well established. But while similar beneficial effects have been described for premature infants, the dropout rate for breastfeeding in families exposed to the uncertainties and stress of the early months of life in the neonatal intensive care unit is very high. The World Health Organization recommends the use of Human Milk Donor Banks to feed infants that cannot be breastfed by their own mothers. These banks are established with the purpose of collecting, screening, processing (including pasteurizing), testing and distributing donated human milk. The potential benefit of donated milk against acute disease elicited by RSV is unknown. The investigators propose to study the role of supplemental donated human milk in the prevention of hospitalizations caused by RSV in non-breastfeeding premature infants. Since the investigators expect the benefits of breast milk to extend beyond protection against RSV, the effect of human milk against respiratory infections elicited by other viruses will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* VLBW preterm neonates (birth weight <1,500 g at birth; gestational age <37 weeks) born alive at any of the two participating maternity hospitals integrating our network in Argentina will be enrolled in the study after signature of informed consent.

Exclusion Criteria:

* VLBW infants older than one month of age (e.g.: transferred from another institution), or formula fed for over ten days, or with congenital heart disease, congenital anomalies of the respiratory tract (i.e.: tracheoesophageal fistula, pulmonary hypoplasia, diaphragmatic hernia), immune suppression, severe malformations affecting breathing (i.e. anencephaly) as well as infants who die prior to completion of the first questionnaire, or living more than 40 km away from the Hospital will be excluded from participation. Infants born from human immunodeficiency virus (HIV) positive mothers will also be excluded

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of respiratory episodes in premature infants | During the first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Fernando P Polack, MD, Principal Investigator — Fundacion Infant
Locations (1):
- Fundacion INFANT, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quigley M, Embleton ND, Meader N, McGuire W. Donor human milk for preventing necrotising enterocolitis in very preterm or very low-birthweight infants. Cochrane Database Syst Rev. 2024 Sep 6;9(9):CD002971. doi: 10.1002/14651858.CD002971.pub6. PMID 39239939